CLINICAL TRIAL: NCT00418223
Title: Detecting Urinary Retention After Child Birth With a Ultrasound Scanner
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Oslo University Hospital, Oslo University Hospital
Other Study IDs: Lukasse-2006; S-06412a
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Urinary Retention
Keywords: Urinary retention; Child birth; Catheterization; Ultrasound
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
The purpose of this study is a systematical registration of ultrasound measurements and urinary volume after catheterization. Based on these pairs of measurements we will calculate the reliability of ultrasound compared with catheter volume.

ELIGIBILITY:
Inclusion Criteria:

* Women with suspected urinary retention

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women after childbirth
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2005-11; Study Completion 2007-02

CONTACTS AND LOCATIONS:
Overall Officials: Leiv A Rosseland, MD, Study Director — Oslo University Hospital
Locations (1):
- Rikshospitalet-Radiumhospitalet HF, Oslo, Norway

REFERENCES:
- [Background] Lukasse M, Cederkvist HR, Rosseland LA. Reliability of an automatic ultrasound system for detecting postpartum urinary retention after vaginal birth. Acta Obstet Gynecol Scand. 2007 Oct;86(10):1251-5. doi: 10.1080/00016340701621478. PMID 17851812